CLINICAL TRIAL: NCT05788653
Title: Comparison of the Effectiveness of Transverse Friction Massage and Thiele Massage in Female Patients With Chronic Pelvic Pain
Brief Title: Comparison of Different Massages Tecniques on Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Sena Öndeş, Principle Investigator, Atlas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SenaOndes1
Record Dates: First submitted 2023-03-10; First posted 2023-03-29 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Chronic Pelvic Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thiele Group (Active Comparator): The group will be given Thiele Massage twice a week for 4 weeks. Thiele massage will be done with a stripping motion in the direction of the pelvic floor muscle fibers. Approximately 15-20 repetitions will be applied to each of the pelvic floor muscle groups for 30 minutes.
  Interventions: Procedure: Thiele Massage
- Transverse Friction Group (Active Comparator): The group will be given Transverse Friction Massage twice a week for 4 weeks. Transverse friction massage will be applied to each tense muscle group and trigger points for 3-5 minutes, crossing the direction of the pelvic floor muscle fibers. Massage duration is approximately 30 minutes for each session.
  Interventions: Procedure: Transverse Friction Massage

INTERVENTIONS:
Procedure: Thiele Massage — Transvaginal Massage
  Arms: Thiele Group
Procedure: Transverse Friction Massage — Transvaginal Massage
  Arms: Transverse Friction Group

SUMMARY:
The aim of this study is to investigate and compare the effectiveness of transverse friction and Thiele massage on pain, quality of life and sexual functions in female patients with chronic pelvic pain. The study will be performed on 20 female patients with pelvic floor muscle tenderness, who applied to the Urology Clinic in Istanbul and were diagnosed with chronic pelvic pain.

ELIGIBILITY:
Inclusion Criteria:

Clinical Diagnosis of Pelvic floor muscle tenderness, Clinical Diagnosis of Chronic Pelvic Pain Syndrome

Exclusion Criteria:

Neurological pathologies ( such as hemiplegia, epilepsy, multiple sclerosis and parkinson's disease) Urogynecological surgery in the last 6 months, Severe pelvic prolapse, Pelvic malignancy and pelvic radiotherapy.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Both intervention methods are transvaginal massage. It can only be applied to female patients.
Enrollment: 20 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 4 weeks
  The Visual Analog Scale is used to determine the severity of pain. At the beginning of a 10 cm long line, there is the phrase "no pain" and "unbearable pain" at the end. The person to be evaluated is asked to put a mark on the scale according to the severity of the pain. Pain intensity is determined by measuring the distance from the expression "No pain" to the area where the person puts a sign. Researchers will take two measurements, at the beginning and at the end of the intervention, to determine the change in pain parameters.
McGill Melzack Pain Questionnaire (MMPQ) | 4 weeks
  The scale consists of four parts. In the first part, the painful place is marked on the human body diagram and it is stated that it is deep and/or superficial. In the second part, where the characteristics of pain are questioned, the words that best describe pain are marked, one from each box out of 20 boxes. In this part, the sensory and perceptual dimensions of pain are evaluated. The third section evaluates the time-dependent variation of pain. In the fourth section, the severity of pain is measured comparatively. The scoring ranges from 0 to 112. A higher score indicates worsening of pain and related parameters. Researchers will take two measurements, at the beginning and at the end of the intervention, to determine the change in pain parameters.
Notthingam Health Profile Questionnaire (NHP) | 4 weeks
  It is a valid and reliable scale that measures general health status in musculoskeletal disorders and chronic diseases. It questions the well-being of individuals in physical, emotional and social areas. The first part consists of 38 questions and six subheadings: pain, emotional reactions, sleep, social isolation, physical activity and energy level. In the second part, it is evaluated to what extent the limitations experienced by individuals in their daily activities due to their health status affect their quality of life. The first part score is calculated between 0-600 points, with a maximum of 100 points for each sub-title, and the second part is calculated between 0-7 points. High scores indicate low quality of life. Researchers will take two measurements, at the beginning and at the end of the intervention, to determine the change in quality of life.
Female Sexual Function Index (FSFI) | 4 weeks
  It is a 5-point Likert-type scale consisting of 19 items and 6 sub-parameters. It evaluates many parameters such as frequency and level of sexual desire, level of arousal, frequency and difficulty of lubrication, ability to maintain lubrication, frequency and difficulty of orgasm, emotional intimacy in sexual intercourse, satisfaction with sexual life, pain during sexual intercourse. The first two questions are calculated between 1-5 points and the other questions between 0-5 points. When the raw scores are multiplied by the coefficients, the highest possible score is 36.0 and the lowest score is 2.0. A high score means that sexual functions are good. The cut-off value of the scale is 26.55. Researchers will take two measurements, at the beginning and at the end of the intervention, to determine the change in female sexual functions.
Bristol Female Lower Urinary System Symptom Index (BFLUSSI) | 4 weeks
  It was developed to evaluate female lower urinary tract symptoms, their severity, and the effects of these symptoms on quality of life and sexual functions. It consists of 34 Likert type questions. 19 questions assess mixing functions, 4 questions assess sexual functions and 11 questions assess quality of life. It consists of 5 sub-parameters, these are storage (questions 1-4), urination (questions 5-7), incontinence (questions 8-12), sexual life (questions 13-14) and quality of life (questions 15-19). Scoring is between 0.71. A high score indicates worsening of lower urinary tract symptoms. Researchers will take two measurements, at the beginning and at the end of the intervention, to determine the change in lower urinary system symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine Hospital, Istanbul, Bağcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided